CLINICAL TRIAL: NCT07105943
Title: Manipulating Exercise Intensity and Affective Responses on a Cardiac Rehabiliattion Program for Patients With Acute Coronary Syndrome: Protocol for a Randomized Controlled Trial
Brief Title: Manipulating Exercise Intensity and Affective Responses for Cardiac Rehabilitation Program Acute Coronary Syndrome Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Collaborators: Universidade Lusófona de Humanidades e Tecnologias (Other); Centro Hospitalar de Leiria (Other); Rede de Investigação em Saúde (Other)
Responsible Party: Principal Investigator, Filipa Januario, Collaborator Member, Instituto Politécnico de Leiria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Instituto Politécnico Leiria
Record Dates: First submitted 2025-07-17; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Affect and Exertion During and Post-exercise
Keywords: acute coronary syndrome; cardiac rehabilitation; physical activity; affective response; motivation
MeSH Terms: conditions — Acute Coronary Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Other: Control
- Experimental (Experimental)
  Interventions: Other: Experimental

INTERVENTIONS:
Other: Control — The intervention will be implemented in the 8 weeks phase 2 cardiac rehabilitation program.
  Both groups will receive a pre-exercise evaluation and 16 individualized training sessions (two per week) based on FITT-VP principles and according to the European Association of Preventive Cardiology (EAPC) guidelines. A complementary physical activity program integrated into their daily life will be prescribed. It will receive regular briefing sessions regarding the health-related benefits of exercise. After these sessions, it will be recommended to maintain physical activity aiming to reach at least 150 min/week of moderate intensity PA.
  Arms: Control
Other: Experimental — As for the experimental group, in the 16 individualized training sessions (two per week), attention will be given to exercise intensity assessment and manipulation, with the goal of optimizing the affective experience of exercise, while also respecting minimum and maximum intensity thresholds as proposed by the EAPC (self-selected intensity within individually defined limits). The pre-exercise evaluation, the number of sessions, and methodological approach will be the same to the control group. In this group it will be presented some awareness of the potential of choosing fun and pleasant activities.
  Arms: Experimental

SUMMARY:
The goal of this clinical trial is to learn if pleasure-oriented exercise intensity manipulation increases physical activity (PA) behavior in patients who have suffered acute coronary syndrome during a cardiac rehabilitation program. The main question it aims to answer is:

• the manipulation of exercise intensity performed to produce more pleasure and arousal will impact the PA behavior? Researchers will compare the PA levels and affective responses to see if the manipulation of exercise intensity guided to pleasure and arousal works to increase PA behavior compared to the control group who will follow a conventional exercise program.

Participants will do:

* sixteen individualized hospital exercise sessions (two per week) and complementary physical activity program integrated into their daily life
* be evaluated before and at the end of the exercise sessions and after 3 months

DETAILED DESCRIPTION:
Ischaemic heart disease remains the top global cause of death, with cases rising by 2.7 million to 9.0 million deaths over the past two decades and between 1990-2019 the percentage of years of life lived with disability increased 83%.

Ischaemic heart disease includes acute coronary syndromes (ACS) that consist of acute myocardial infarction (AMI) and unstable angina. After ACS there is a greater risk of recurrence of the event, arrhythmias, heart failure and sudden death. These patients also have a lower quality of life which impacts their physical function and psychological well-being. ACS represent a substantial direct cost and economic burden for national health systems. Prevention must be prioritized and the emphasis on encouraging physical activity (PA) and routine exercise has become more vital than ever.

The 2023 European Society of Cardiology Guidelines for the management of ACS recommend that all patients participate in a medically supervised, structured, comprehensive cardiac rehabilitation (CR) program with a multidisciplinary team. Its core components are patient assessment, management and control of cardiovascular risk factors, PA counselling, prescription of exercise training, dietary advice, tobacco counselling, patient education, psychosocial management, and vocational support. Exercise plays a key role having a Class I, Level A evidence supporting its benefits, while specific components such as aerobic PA and muscle-strengthening exercises are supported by Class I, Level B evidence. CR plays a crucial role in lowering rates of hospitalization, fatal and non-fatal myocardial infartion, while improving exercise capacity and quality of life. There is also a reduction in healthcare costs for participants in a CR program compared with nonparticipants.

CR typically consists of three phases: phase 1 (in-hospital), phase 2 (mostly in an outpatient setting: centre-based or home-based) and phase 3 (maintenance phase in outpatient or community settings, aimed at sustaining lifestyle changes). Phase 2 CR is typically provided as an outpatient program, lasting between 8 to 24 weeks, with sessions offered 3 to 7 days per week.

A progressive program of structured exercise and PA are a fundamental part of a CR program. Exercise training should be tailored to the individual, following a thorough clinical assessment that includes risk stratification, behavioral traits, personal objectives, and exercise preferences. Exercise should be prescribed based on FITT-VP (frequency, intensity, time, type of exercise, volume, and progression) model. It is recommended to do aerobic training at a frequency of at least 3 days per week, with a preference for 6-7 days per week, at a moderate or moderate-to-high intensity. It is also advised to do resistance training, 2 days per week, at 30-70% of one-repetition maximum (1RM) for the upper body and 40-80% of 1RM for the lower body, with 12-15 repetitions/set. After the end of the CR program (i.e., beginning of phase 3), ACS patients should accumulate at least 30 minutes per day, 5 days per week of moderate intensity PA (equating to 150 minutes per week) or 15 minutes per day, 5 days per week of vigorous intensity PA (equating to 75 minutes per week), or a combination of both. These PA levels are needed for reducing disease progression and increasing quality of life.

Despite being aware of the benefits of regular PA and intending to stay active, many patients struggle to adopt or maintain these behaviors in the long-term. One-third of their sample did not reach the recommended PA levels in the first weeks after discharge from CR. Moreover, in long-term approximately 66% of patients failed to meet the established PA goal.

The central problem is the sustainability of PA after phase 2 CR. Therefore, strategies aimed at improving patients' attitudes toward and adherence to exercise are warranted.

Patient should be actively participating in their exercise program, tailoring it to their needs and preferences, as personalized care increases the likelihood of improved adherence to an exercise routine during and after CR. Knowing that adherence is influenced by complex psychological factors, exploring them should be a crucial effort in such programs. As such, exploring the individual motivation may be a relevant consideration for such effort.

Patient should be actively participating in their exercise program, tailoring it to their needs and preferences, as personalized care increases the likelihood of improved adherence to an exercise routine during and after CR. Knowing that adherence is influenced by complex psychological factors, exploring them should be a crucial effort in such programs. As such, exploring the individual motivation may be a relevant consideration for such effort.

Improving adherence to phase 3 CR recommendations The success of a CR program could be measured by the extent of the individual recovery process and the ability to introduce sustainable, long-lasting behavioral changes capable of preventing relapse, where PA is a crucial component. In apparently healthy individuals, several theories and approaches have been used for adherence support and healthy habits adoption. These are often grounded in motivational aspects, where several prominent theories have been used.

In the CR context, some efforts have been made for this purpose. Some studies used Self-Determination Theory assumptions to explore its potential role in supporting PA in these patients. Results indicated that promoting basic psychological needs satisfaction and supporting autonomy predicted PA/exercise behavior. In other studies, the Theory of Planned Behavior was used as the theoretical background for the same exploration, and once again, evidence was found to the theory underpinnings, mainly for intention, and their positive relation to PA. These are just a few examples of how the study of motivation has been used in the past in CR programmes to try to improve patient adherence in later phases and to support lifestyle changes. However, these are also examples that mimic several of the current issues in translating motivational and behavioral theories into practice, not only in these programmes, but also for general PA promotion. For once, these suggestions emerge from cross-sectional and longitudinal studies, thus evidencing the struggle that translating and operationalization the distinct theories' assumptions brings, given the absence in the last decades of experimental efforts in the most of contexts. Then, it is also possible to easily verify that CR programmes still struggle to improve PA adherence in later stages of the recovery process, even though the unquestionable, evidence-based indication of its worthiness, and the ever-growing support emerging from psychological theories of motivation.

Given that this is not an exclusive problem in this context and patients, researchers concerned with the motivational aspects of PA have been exploring other possibilities and approaches. One that will be used to support the current study's experimental approach is grounded on the emerging line of the psychological study of affectivism. This line of thought assumes that non-rational aspects of behavior, as is the case with core affect, can influence individual motivational development through a hedonistic lens (i.e., tendency to approach activities that promote pleasurable sensations, and to avoid those experienced as unpleasant ones). Core affect is posited to be a neurophysiological state that is consciously accessible as a simple, nonreflective feeling that is an integral blend of hedonic (pleasure-displeasure) and arousal (sleepy-activated) values. Some recent efforts grounded on dual-process theories, where core affect is an integral component of implicit and, indirectly, reflective pathways, have been made in similar CR programmes. That showed support for the role of affective attitudes in supporting PA, thus evidencing the emerging concern and focus of potential affective constructs in this matter.

Current study In PA settings, several conditions can manifest in these feelings (i.e., core affect) and thus impact motivation, but one stands as the one more directly responsible - exercise intensity. As posited by the Affect and Health Behavior Framework (AHBF) and the Dual Mode Theory (DMT), intensity is closely related to core affect manifestations. Generally, the exposure to higher intensities is tendentially experienced as unpleasant, and lower intensities as pleasant. Often, a pleasurable heterogeneity zone emerges between some metabolic (e,g., ventilatory threshold) or load (~75% RM) thresholds that anticipate the decrease and often emergence of unpleasant responses . A successful and individual experience of pleasurable responses is posited to support motivation development and subsequently align with being physically active and supporting lifestyle changes, but experimental efforts to test these theoretical assumptions are lacking.

There is a study where it was manipulated the exercise intensity to promote pleasurable experiences in individualized exercise sessions in fitness centers. An 8-week follow-up showed that the experimental group had a 77% higher session attendance when compared to the control group (14.35 vs. 8.13). This was achieved using the ACSM exercise guidelines for healthy adults, were the exercise intensity, in the experimental group, was adjusted to support pleasurable affective responses and align with individual intensity preference and tolerance, in an autonomy supportive manner.

The current study will be developed in an ongoing CR program aligned with the European Association of Preventive Cardiology (EAPC) guidelines, which presents its own specification of the FITT-VP principles. As such, the general conditions to allow the manipulation of exercise intensity and the replication of the motivational approach are present and are inherently of relevance for increasing phase 2 and 3 CR physical activity levels.

ELIGIBILITY:
Selection criteria include:

* patients older than 18 years
* diagnosis of ACS within the past 12 months who have not previously participated in a CR program
* patients classified as low-risk (Class B) according to the American Heart Association: (a) New York Heart Association (NYHA) class I or II, (b) exercise capacity greater than 6 METs, (c) no evidence of heart failure, (d) no signs of myocardial ischemia or angina at rest or during exercise testing at or below 6 METs, (e) appropriate systolic blood pressure response during exercise, and (f) absence of sustained or non-sustained ventricular tachycardia at rest or during exercise.

Standard exclusion criteria include:

* left ventricular ejection fraction (LVEF) < 40% at rest
* uncontrolled arrythmias (e.g., complex ventricular arrhythmias, atrial fibrillation or flutter with rapid ventricular response, second-degree atrioventricular block Mobitz type II, or third-degree atrioventricular block)
* presence of an implantable cardiac device
* symptomatic peripheral arterial disease
* comorbidities that may interfere with the ability to perform the exercise program safely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Physical activity levels by International Physical Activity Questionnaire - Short Form | At baseline (the week before phase 2 cardiac rehabilitation program), end of the intervention (first week after the intervention) and at 3 months after it
  International Physical Activity Questionnaire - Short Form: physical activity will be assessed by a continuous variable, expressed in MET-minutes per week. It will be applied in order to evaluate the same week of accelerometry.
Affective responses in exercise sessions phase 2 cardiac rehabilitation program - Felt Arousal Scale | During all exercise sessions (twice a week for 8 weeks) will be administered at 10-min intervals during the aerobic activity; immediately after the fourth and eighth resistance exercises set and in the last 15 sec of the set of the fifth stretch exercise
  Felt Arousal Scale is a 6-point scale ranging from 1 ("Low arousal") to 6 ("High arousal") that assesses perceived activation
Physical activity levels by accelerometry | At baseline (the week before phase 2 cardiac rehabilitation program), end of the intervention (first week after the intervention) and at 3 months after it
  We will use the ActiGraph® GT3X+ (Pensacola, FL) accelerometer. The researcher will distribute the accelerometers to all participants, that will be instructed to wear the device on an elastic belt around their waist on the right side for seven consecutive days, taking it off only for water-based activities (e.g., shower and swimming) and sleep. Participants will be asked to carry out their usual activities during data collection. The cut points and wear time validation criteria will be used to define the time spent in each intensity period and to define a valid register. A day will be considered valid with at least 600 minutes of use, and each participant will have to present at least four valid days, including a at least one weekend day to be included in the analysis. Compliance with PA recommendations for public health will be assessed according to EAPC recommendations (150 min/week of MVPA defined as ≥ 21.4 min/day).
Affective responses in exercise sessions phase 2 cardiac rehabilitation program - Feeling Scale | During all exercise sessions (twice a week for 8 weeks) will be administered at 10-min intervals during the aerobic activity; immediately after the fourth and eighth resistance exercises set and in the last 15 sec of the set of the fifth stretch exercise
  Feeling Scale is an 11-point scale ranging from -5 ("Very bad") to +5 ("Very good"), which assesses the affective valence (how one feels at that given moment)

SECONDARY OUTCOMES:
Participation in the complementary physical activity program | In the 8 weeks of the intervention
  minutes-week of physical activity
Anticipated affective response | 5 minutes before the exercise sessions 1, 8 and 16 during the intervention (exercise sessions are twice a week for 8 weeks)
  Anticipated affective response to a future exercise session measured with the adaptation of the Empirical Valence Scale will be used to assess anticipated affective response to exercise sessions. This instrument uses 15 empirically spaced verbal anchors ranging from -100 ("Most unpleasant imaginable") to +100 ("Most pleasant imaginable"). Participants will respond to the question "Considering the workout you are about to begin (previously explained/remembered), how do you think it will make you feel?".
Final remembered affect to the previous exercise session | 5 minutes after exercise sessions 1, 8 and 16 during intervention (exercise sessions are twice a week for 8 weeks)
  Remembered affect of previous exercise session measured with the Visual Analog Scale A Visual Analog Scale (VAS) will be used to assess remembered exercise pleasure/displeasure. Participants will be asked to rate "How did your last workout make you feel?". This scales ranges from +100 ("very pleasant") to -100 ("very unpleasant").
Intention to continue exercising | 5 min before session 1 and 5 min after session 16 during intervention (exercise sessions are twice a week for 8 weeks). At the end of the intervention (first week after the intervention) and at 3 months after it
  The behavioral intention will be assessed using three items (e.g., "I will continue to practice physical exercise in the next 6 months as I recently practiced [with or without personal trainer] or in a very similar way (same type, frequency, duration, and intensity"). Responses are entered using a 7-point ordinal scale ranging from 1 ("Absolutely not") to 7 ("Absolutely yes").
Exercise habit | 5 min before session 1 and 5 min after session 16 during intervention (exercise sessions are twice a week for 8 weeks). At the end of the intervention (first week after the intervention) and at 3 months after it
  The Self-Report Behavioral Automaticity Index will be used to assess behavioral habit development. The instrument consists of four items (e.g., "I do without thinking") answered on a 7-point Likert scale, ranging from 1 ("Totally disagree") to 7 ("Totally agree").
Exercise enjoyment | 5 minutes before session 1 and 5 minutes after sessions 8 and 16 during intervention (exercise sessions are twice a week for 8 weeks).
  Exercise enjoyment measured with the the Physical Activity Enjoyment Scale (PACES). This questionnaire includes eighteen items related to "how do you felt during the exercise you have recently completed?" that are answered using a 7-point bipolar scale with antithetical statements (e.g., item 1: "I loved it - I hated it").
Intensity preference, tolerance, and agreement of exercise | 5 minutes before session 1 and 5 minutes after session 8 and 16 during intervention (exercise sessions are twice a week for 8 weeks).
  The Preference for and Tolerance of Exercise Intensity Questionnaire (PRETIE-Q) will be used to assess individual differences in intensity-preference, intensity-tolerance, and the agreement between self-reported preference and tolerance with the intensity experienced during the preceding exercise session. The instrument is composed of 10 items (five for each factor; preference: "Low-intensity exercise is boring"; tolerance: "Feeling tired during exercise is my signal to slow down or stop") answered on a 5-point Likert scale ranging from 1 ("Totally disagree") to 5 ("Totally agree"). The two additional questions proposed by this instrument version to assess agreement will also be used as recommended.
Motivation to exercise | 5 minutes before session 1 and 5 minutes after session 8 and 16 during intervention (exercise sessions are twice a week for 8 weeks).
  Intrinsic motivation from the the Intrinsic Motivation Inventory will be used. Minor adaptations to the wording will be made to ensure relevance to the context of exercise (e.g., vs. sport) following the example of adaptations in similar studies . For example, "I am satisfied with my performance at this task" (perceived competence) will be adapted to "I am satisfied with my performance in these workouts".
Autonomy in exercise practice | 5 minutes before session 1 and 5 minutes after session 8 and 16 during intervention (exercise sessions are twice a week for 8 weeks).
  Autonomy in exercise practice measured with the perceived choice scale of the Intrinsic Motivation Inventory. Minor adaptations to the wording will be made to ensure relevance to the context of exercise (e.g., vs. sport) following the example of adaptations in similar studies . For example, "I believe I had some choice about doing this activity" (perceived choice) will be adapted to "I believe I had some choice during these workouts". One item will be added to the perceived choice subscale regarding the freedom to select exercise intensity, i.e., "I felt I had the choice to switch the intensity of exercise as I wished".
Abdominal Circumference | Baseline, at the end of the intervention (first week after the intervention) and at 3 months after it
  The measurement will be taken with the patient standing, naked on the upper part, the measuring tape is placed at the midpoint between the costal margin and the upper edge of the iliac crest, at the end of expiration, with the measuring tape straight and without tightening
Body mass index (BMI) | Baseline, at the end of the intervention (first week after the intervention) and at 3 months after it
  BMI (weight (kg) / [height (m)]²).
Body weight | Baseline, at the end of the intervention (first week after the intervention) and at 3 months after it
  Body weight (kg) will be measured using an electronic balance.
Height | Baseline
  Height (m) will be obtained from identification cards

OTHER OUTCOMES:
Resting blood pressure | Before and after all exercise sessions during the intervention (exercise sessions are twice a week for 8 weeks).
  Resting blood pressure (mmHg) - systolic and diastolic. It will be tested on the right upper limb of the seated patient.
Heart rate during exercise | During all the exercise sessions during the intervention (exercise sessions are twice a week for 8 weeks).
  Heart rate will be monitored using a telemetry system
Perceptions of effort | During all exercise sessions the Borg Scale will be administered at 10-min intervals during the aerobic activity; immediately after the set of the fourth and eighth resistance exercises, and in the last 15 sec of the fifth stretch exercise
  Perceptions of effort assessed by Borg Rating of Perceived Exertion Scale 15-point (Borg Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade Local de Saúde da Região de Leiria, Leiria, Portugal

IPD SHARING:
Plan to Share IPD: No